CLINICAL TRIAL: NCT05699746
Title: A Randomized Controlled Trial of CAPEOX vs Observation in Early-stage Colorectal Cancer Patients With Positive MRD After Curative Surgery
Brief Title: CAPEOX vs Observation in Colorectal Cancer Patients With Positive MRD
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Zhejiang University (Other)
Collaborators: GeneCast Biotechnology Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Ding Ke-Feng, Professor, Zhejiang University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IR2022577
Record Dates: First submitted 2023-01-16; First posted 2023-01-26 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Capecitabine; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CAPEOX (Experimental): Drug CAPEOX (Oxaliplatin 130 mg/m2 IV day 1, Capecitabine 1000 mg/m2, twice daily PO for 14 days, repeat every 3 weeks) for at most 8 cycles.
  Interventions: Drug: Capecitabine tablets; Drug: Oxaliplatin
- Observation (No Intervention): Patients undergo active surveillance

INTERVENTIONS:
Drug: Capecitabine tablets — Capecitabine 1000 mg/m2, twice daily PO for 14 days, repeat every 3 weeks, for at most 8 cycles.
  Arms: CAPEOX
Drug: Oxaliplatin — Oxaliplatin 130 mg/m2 IV day 1, combined with Capecitabine, for at most 8 cycles.
  Arms: CAPEOX

SUMMARY:
Patients with stage Ⅰ colorectal cancer or stage Ⅱ colon cancer usually have a good prognosis and are not recommended to receive adjuvant chemotherapy after radical surgery. With the advances in liquid biopsy technology, detection of circulating tumor DNA (ctDNA) can effectively identify early-stage cancer patients with minimal residual disease (MRD) after surgery. According to the growing number of MRD studies in solid tumor, colorectal cancer patients with ctDNA-MRD detection have a poor clinical outcome and are likely to relapse within two years. This study aims to assess the efficacy of adjuvant chemotherapy with capecitabine plus oxaliplatin (CAPEOX) compared with conventional observation in MRD-positive patients with stage I colorectal cancer and clinically low-risk stage II colon cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Colorectal cancer confirmed by pathology, and the TNM stage (AJCC v8) is stage I or stage II. Stage II patients have T3 colonic adenocarcinoma with proficient mismatch-repair system (by immunohistochemistry for four mismatch repair proteins MSH1, MSH2, MSH6, and PMS2) and have no the following clinical risk factors: a) less than 12 lymph nodes examined; b) mucinous carcinoma; c) poor differentiation; d) bowel obstruction or perforation; e) lymphatic/vascular invasion, perineural invasion; f) close, indeterminate, uncertain, positive margins
2. ECOG performance status 0-1
3. No neoadjuvant therapy before surgery
4. Appropriate for active surveillance (i.e., no adjuvant chemotherapy) based on current practice patterns or according to the Chinese Society of Clinical Oncology guidelines for Colorectal Cancer (version 2022)
5. No history of other primary cancers in the past 3 years
6. No history of bone marrow, stem cell or organ transplant
7. Blood samples from 7 to 21 days after surgery were tested positive for ctDNA (tested by MinerVa MRD assay)
8. Pregnancy test done within 14 days before randomization must be negative (for women of childbearing potential only)
9. Voluntarily join the study and sign the informed consent document
10. No unstable or any medical condition that affects patient safety and study compliance evaluated by researchers
11. Availability and provision of adequate surgical tumor tissue for molecular diagnostics

Exclusion Criteria:

1. Patients with multiple primary colorectal cancers
2. Patients with another primary cancer
3. Patients have the following conditions by blood test, or have obvious contraindication in adjuvant chemotherapy:

   1. Moderate/severe renal impairment (GFR<30 ml/min), as calculated by the Cockcroft and Gault equation
   2. Absolute neutrophil count <1.5×109/L
   3. Platelet count < 75×109/L
   4. Hemoglobin <90 g/L
   5. Aspartate aminotransferase/Alanine aminotransferase >2.5 × upper limit of normal
4. Lactating women
5. Have serious or uncontrolled medical condition that may preclude compliance with the protocol

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2023-03 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Recurrence-free survival | 18 months

SECONDARY OUTCOMES:
Clearance of circulating tumor DNA (ctDNA) | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Kefeng Ding, MD, PhD, Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (4):
- China (4):
  - Changhai Hospital of Shanghai, Shanghai, Shanghai Municipality
  - Sir Run Run Shaw Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Second Affiliated Hospital Zhejiang University College of Medicine, Hangzhou, Zhejiang
  - The second hospital of Ningbo City, Ningbo, Zhejiang

IPD SHARING:
Plan to Share IPD: No